CLINICAL TRIAL: NCT05726097
Title: Optimization of the Bowel Preparation Regimen for Colon Capsule Endoscopy Procedure
Brief Title: Bowel Preparation Regimen for Colon Capsule Endoscopy Procedure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022-06303-02
Record Dates: First submitted 2022-12-22; First posted 2023-02-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer; Inflammatory Bowel Diseases; Gastrointestinal Bleed; Colon Polyp
Keywords: colon capsule endoscopy; panenteric capsule endoscopy; colon preparation
MeSH Terms: conditions — Colonic Neoplasms; Inflammatory Bowel Diseases; Gastrointestinal Hemorrhage; Colonic Polyps | interventions — Polyethylene Glycols; sodium phosphate; Ascorbic Acid; Diatrizoate Meglumine; picosulfate sodium; prucalopride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard preparation regimen (Active Comparator): 4 L polyethylene glycol as laxative 30 + 15 mL sodium phosphate as a booster
  Interventions: Drug: polyethylene glycol; Drug: sodium phosphate
- Optimized preparation regimen (Experimental): 1 L polyethylene glycol + ascorbic acid as laxative and gastrografin and magnesiumoxid + sodium picosulfate as a booster
  Interventions: Drug: polyethylene glycol + ascorbic acid; Drug: gastrografin; Drug: magnesiumoxid + sodium picosulfate
- Optimized preparation regimen with prucalopride (Experimental): 1 L polyethylene glycol + ascorbic acid as laxative and gastrografin and magnesiumoxid + sodium picosulfate as a booster + 2 mg of prucalopride
  Interventions: Drug: polyethylene glycol + ascorbic acid; Drug: gastrografin; Drug: magnesiumoxid + sodium picosulfate; Drug: prucalopride

INTERVENTIONS:
Drug: polyethylene glycol — colonic preparation
  Other Names: Laxabon
  Arms: Standard preparation regimen
Drug: sodium phosphate — colonic preparation
  Other Names: Phosphoral
  Arms: Standard preparation regimen
Drug: polyethylene glycol + ascorbic acid — colonic preparation
  Other Names: Plenvu
  Arms: Optimized preparation regimen; Optimized preparation regimen with prucalopride
Drug: gastrografin — colonic preparation
  Arms: Optimized preparation regimen; Optimized preparation regimen with prucalopride
Drug: magnesiumoxid + sodium picosulfate — colonic preparation
  Other Names: Picoprep
  Arms: Optimized preparation regimen; Optimized preparation regimen with prucalopride
Drug: prucalopride — colonic preparation
  Other Names: Resolol
  Arms: Optimized preparation regimen with prucalopride

SUMMARY:
The study aims to investigate the effect of the optimized bowel preparation and boost regimens on colon capsule endoscopy procedures, specifically on cleanliness and completion rate.

DETAILED DESCRIPTION:
Colon capsule endoscopy (CCE) is a promising modality for lower gastrointestinal (GI) investigations in clinical routine and screening. Furthermore, the double-headed camera capsules are being applied for panenteric investigations, with promising results. The major limitation to its use has been finding a bowel preparation that will clean the colon adequately for good visualization of the mucosa and help propel the capsule using boosters through the colon. To achieve wider CCE adoption, challenges regarding completion rates (CR) and adequate cleanliness rates (ACR) must be handled. CR and ACR should be improved to meet the standards for optical colonoscopy (OC) from the European Society of GI Endoscopy (ESGE). ESGE recommends both CR and ACR ≥ 90%. Recently, a meta-analysis of preparation regimens for CCE confirmed that CR and ACR were suboptimal.

This study is designed to investigate the CR, ACR, and diagnostic yield (DY) of very low-volume polyethylene glycol (PEG) - based laxative compared to a conventional high-volume laxative and the use of different boosters.

All consecutive patients referred for colon capsule endoscopy will be enrolled in the study. PillCam® Crohn's capsule will be used. Patients will undergo a split-dose bowel preparation with a very low-volume PEG-based laxative. In the study arm nr1 gastrografin and magnesiumoxid + sodium picosulfate will be used. In the study arm Nr 2, the same regimen will be used but completed with 2 mg of prucalopride before ingesting the capsule. The results of the study arms will be compared to the previously used standard regimen with 4 L of PEG as a laxative and sodium phosphate as a booster.

The images from the colon capsule will be reviewed, and the quality of bowel preparation (cleanliness rates) and completion rate will be evaluated. Patient tolerance of the bowel preparations and diagnostic yield of colon capsule endoscopy using the different preparation regimens will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject referred for clinical colon/panenteric examination
* Subject received an explanation about the nature of the study and agreed to provide written informed consent

Exclusion Criteria:

* Subject with dysphagia or any swallowing disorder
* Subject with a prior stomach, small bowel, or colonic resection
* Subject with severe renal insufficiency
* Subject with any allergy or other known contraindication to the medications used in the study
* Women who are either pregnant or nursing
* Subject suffers from life threatening conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Completeness rate | Within 3 months after completed capsule colonoscopy
  Visualization of the hemorrhoidal plexus or an excreted capsule
Adequate cleanliness rate | Within 3 months after completed capsule colonoscopy
  Assessment of the quality of the bowel preparation using a the 4-point Leighton-Rex scale

SECONDARY OUTCOMES:
Transit times | Within 3 months after completed capsule colonoscopy
  Determining the amount of time for the capsule to transit through the stomach, small bowel and large bowel for the different preparations
Diagnostic yield | Within 3 months after completed capsule colonoscopy
  Findings in the small and large bowel
Assessment of patient tolerance of the bowel preparations | Within 3 months after completed capsule colonoscopy
  Survey questionnaire to be completed by participants at the time of the colon capsule endoscopy assessing the tolerability of the preparation and side effects

CONTACTS AND LOCATIONS:
Overall Officials: Ervin Toth, MD PhD, Principal Investigator — Department of Gastroenterology, Skåne University Hospital, Malmö, Lund University, Sweden
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05726097/Prot_SAP_ICF_000.pdf